CLINICAL TRIAL: NCT03126838
Title: Diaphragmatic Dysfunction and Cardiac Surgery; Perioperative Assessment and Effect on Outcome; Prospective Observational Study
Brief Title: Diaphragmatic Dysfunction and Cardiac Surgery; Perioperative Assessment and Effect on Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Institute, Egypt (Other Government)
Responsible Party: Principal Investigator, Ibrahim Shawky Morsy Omara, 32 family housing, area 8, El obour city, Qalubia, Egypt, National Heart Institute, Egypt
Other Study IDs: NHIEgypt ,670/2017
Record Dates: First submitted 2017-03-11; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Diaphragm Disease
Keywords: diaphragm; ultrasound; dysfunction; cardiac surgery; weaning

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diaphragmatic dysfunction: diaphragmatic displacement < 10 ml, and / OR diaphragmatic thickening fraction < 36 %.
- non diaphragmatic dysfunction: diaphragmatic displacement > 10 ml, and / OR diaphragmatic thickening fraction > 36 %.

SUMMARY:
This study evaluates incidence of diaphragmatic dysfunction after cardiac surgery and its effect on outcome of surgery.

DETAILED DESCRIPTION:
Diaphragmatic dysfunction will be assessed by ultrasonography the day before operation and first post operative day, by measuring diaphragmatic thickening during inspiration and expiration.incidence of diaphragmatic dysfunction and its effect on outcome of surgery then will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* Planned cardiac surgery
* Ready for weaning from mechanical ventilation (fraction of inspired oxygen (FIO2) ≤ 50%, positive end-expiratory pressure(PEEP) level≤ 5 centimeter water (cmH2O), respiratory rate ≤30 breaths/min, partial pressure of oxygen in arterial blood(PaO2)/FIO2 ratio >200 , Glasgow coma score ≥14).
* Stable cardiovascular status (i.e., heart rate <120 beats/min; systolic blood pressure, 90-160 mmHg; and no or minimal vasopressor use, i.e., dopamine or dobutamine ≤5 μg/kg/min or noradrenaline ≤0.05 μg/kg/min).
* Stable metabolic status (i.e., electrolytes and glycaemia within normal range, body temperature <38 °C, hemoglobinemia ≥8-10 g/dL).

Exclusion Criteria:

* Patients with a history of diaphragmatic or neuromuscular disease or evidence of pneumothorax or pneumomediastinum.
* Patients with low EF (EF ≤ 30%).
* Patients with post-operative cerebrovascular stroke.
* Reventilation due to cardiac cause ( arrest, arrhythmias, or failure)
* Patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 adult patients who are ready for elective cardiac surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic excursion. | at the beginning of the spontaneous breathing trial (around 4hours after surgery).
  diaphragmatic excursion (displacement, cm)
diaphragmatic dysfunction post cardiac surgery. | at the beginning of the spontaneous breathing trial (around 4hours after surgery).
  diaphragmatic thickening fraction [Thickness at end inspiration - Thickness at end expiration]
  / Thickness at end expiration

SECONDARY OUTCOMES:
. Diaphragmatic excursion | the day before surgery
  diaphragmatic excursion (displacement, cm)
• Diaphragm dysfunction before surgery | the day before surgery
  diaphragmatic thickening fraction [Thickness at end inspiration - Thickness at end expiration]
  / Thickness at end expiration
Left ventricular ejection fraction | the day before surgery
  as indicator of cardiac function
• Total ventilation time | from time of addmission to surgical ICU up to 1 week
  in term of hours (in diaphragmatic dysfunction group)
• Extracorporeal circulation duration | peroperative
  cardiopulmonary bypass time in term of minutes
• Ventilation free days. | from time of admission to surgical ICU up to 1 week
  after extubation first time tell end of ICU stay, in term of days (in diaphragmatic dysfunction group)
• Total ICU stay | from time of admission to surgical ICU up to 1 week
  in term of days (in diaphragmatic dysfunction group)

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Institute, Giza, Embaba, Egypt

IPD SHARING:
Plan to Share IPD: No